CLINICAL TRIAL: NCT03977779
Title: Prospective Evaluation of the Use of a Biodegradable Endoprothesis in the Prevention of Post-Endoscopic Retrograde CholoangioPancreatography Pancreatitis
Brief Title: Evaluation of the Use of a Biodegradable Endoprothesis in the Prevention of Post-Endoscopic Retrograde CholoangioPancreatography Pancreatitis
Acronym: ARCHIMEDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ARCHIMEDE-PANCREAS-IPC
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Jaundice; Biliary Stricture; Sphincter of Oddi Dysfunction
Keywords: biodegradable stent; Post-Endoscopic Retrograde CholoangioPancreatography Pancreatitis
MeSH Terms: conditions — Jaundice, Obstructive; Sphincter of Oddi Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prophylactic biodegradable pancreatic stent placement (Experimental)
  Interventions: Device: Placement of ARCHIMEDES fast biodegradable stent during the Endoscopic Retrograde CholoangioPancreatography

INTERVENTIONS:
Device: Placement of ARCHIMEDES fast biodegradable stent during the Endoscopic Retrograde CholoangioPancreatography — The ARCHIMEDES Fast biodegradable pancreatic stent will be placed during the Endoscopic Retrograde CholoangioPancreatography

SUMMARY:
The use of an endoprothesis in a pancreatic duct is a measure to minimize the incidence and severity of Post-Endoscopic Retrograde CholoangioPancreatography Pancreatitis. In this study we will evaluate the use of a Biodegradable Endoprothesis: Archimede Fast Biodegradable Pancreatic Stent in patients with high risk of Post-Endoscopic Retrograde CholoangioPancreatography Pancreatitis.The ARCHIMEDES Fast biodegradable pancreatic stent will be placed during the Endoscopic Retrograde CholoangioPancreatography. The efficacy and the security of the device will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Patients at risk of developing a Post-Endoscopic Retrograde CholoangioPancreatography Pancreatitis (procedure and/or patient-related risk factors

Exclusion Criteria:

* Pregnant or breastfeeding women
* Recent diagnosis (<1 month) of acute pancreatitis
* contraindication to endoscopy
* Hypersensitivity to indomethacine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a complete clearance of the biodegradable stent | Day 15
  The degradation of the stent will be evaluated both duodenoscopy/fluoroscopy and endoscopy 15 days after its placement

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region, France